CLINICAL TRIAL: NCT01574417
Title: The Effects of Plant Stanol Esters on Intestinal Mucosal Gene Expression Profiles and Microbiota Composition in Healthy Human Subjects
Brief Title: Plant Stanols and Gene Expression Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Raisio Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC 12-3-005
Record Dates: First submitted 2012-03-20; First posted 2012-04-10 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Hypercholesterolemia
Keywords: Plant stanols; Gene expression profile; Microbiota
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plant stanol-enriched margarine (Experimental)
  Interventions: Dietary Supplement: plant stanol-enriched margarine
- control margarine (Placebo Comparator)
  Interventions: Dietary Supplement: control margarine

INTERVENTIONS:
Dietary Supplement: control margarine — Subjects will undergo a postprandial test for 5.5 hours, in which 26.7gram of the control margarine is consumed together with a high-fat milkshake.
  Daily consumption of 20 gram of a control margarine (providing daily 3.0 gram of plant stanols), for a period of 3 weeks.
  Arms: control margarine
Dietary Supplement: plant stanol-enriched margarine — Subjects will undergo a postprandial test for 5.5 hours, in which 26.7gram of the plant stanol-enriched margarine is consumed together with a high-fat milkshake.
  Daily consumption of 20 gram of a plant stanol-enriched margarine (providing daily 3.0 gram of plant stanols), for a period of 3 weeks.
  Arms: Plant stanol-enriched margarine

SUMMARY:
Plant sterols and stanols are dietary components that are naturally present in plants. Their biological function in plants is comparable with these of cholesterol in animals. They are structurally related to cholesterol, but are absorbed by enterocytes to a much lesser extent. It is generally accepted that they inhibit intestinal cholesterol absorption and consequently lower serum low-density lipoprotein (LDL) cholesterol concentrations up to 10% at daily intakes of 2.5 g. The exact underlying mechanism of the plant sterol/stanol mediated reduction in intestinal cholesterol absorption is still unknown. It has been suggested that they lower the activity of sterol uptake transporters like Niemann-Pick C1 like 1 protein (NPC1L1) in enterocytes, otherwise several studies indicated that these compounds could activate the liver X receptor (LXR) in enterocytes, thereby activating the ABC transporters involved in the intestinal cholesterol metabolism, whereas recently suggestions have been made that plant sterols and stanols activate transintestinal cholesterol excretion (TICE). This is the direct cholesterol secretion from the blood into the intestinal lumen, in which the enterocytes play a central role. None of these assumptions have so far been evaluated in humans.

Objective: The major objective of the present study is to examine the acute effects of dietary plant stanol esters on the intestinal mucosal gene expression profiles in intestinal biopsies in healthy volunteers. The minor objective is to investigate whether semi-long-term use (3 weeks) of plant stanol esters have an effect on microbiota composition.

DETAILED DESCRIPTION:
lant sterols and stanols are dietary components that are naturally present in plants. Their biological function in plants is comparable with these of cholesterol in animals. They are structurally related to cholesterol, but are absorbed by enterocytes to a much lesser extent. It is generally accepted that they inhibit intestinal cholesterol absorption and consequently lower serum low-density lipoprotein (LDL) cholesterol concentrations up to 10% at daily intakes of 2.5 g. The exact underlying mechanism of the plant sterol/stanol mediated reduction in intestinal cholesterol absorption is still unknown. It has been suggested that they lower the activity of sterol uptake transporters like Niemann-Pick C1 like 1 protein (NPC1L1) in enterocytes, otherwise several studies indicated that these compounds could activate the liver X receptor (LXR) in enterocytes, thereby activating the ABC transporters involved in the intestinal cholesterol metabolism, whereas recently suggestions have been made that plant sterols and stanols activate transintestinal cholesterol excretion (TICE). This is the direct cholesterol secretion from the blood into the intestinal lumen, in which the enterocytes play a central role. None of these assumptions have so far been evaluated in humans.

Objective: The major objective of the present study is to examine the acute effects of dietary plant stanol esters on the intestinal mucosal gene expression profiles in intestinal biopsies in healthy volunteers. The minor objective is to investigate whether semi-long-term use (3 weeks) of plant stanol esters have an effect on microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-60 years
* BMI between 20-30kg/m2
* mean serum total cholesterol < 7.8mmol/L

Exclusion Criteria:

* unstable body weight
* active cardiovascular diseases
* gastrointestinal diseases
* use of cholesterol-lowering drugs
* use of lipid-lowering therapy
* abuse of drug or alcohol
* pregnant or breast-feeding women
* current smoker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
intestinal mucosal gene expression profiles | Measured at day 8 and day 64. Changes will be calculated between day 8 and day 64.

SECONDARY OUTCOMES:
microbiota composition | measured after 3 weeks consumption of controle margarine and the plant stanol-enriched margarine. Changes will be calculated between these 2 interventions.
lipoprotein profile | measured at baseline and after 3 weeks
plasma glucose concentration | measured at day 8 and day 64, on 8 time points
plasma plant stanol concentration | measured at baseline and after 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jogchum Plat, Dr, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands